CLINICAL TRIAL: NCT01405690
Title: A Pilot Study: The Role Of Noninvasive 320-Row Multidetector Computer Tomography Coronary Angiogram In Predicting Perioperative Cardiac Complications In Patients Referred For Noncardiac Surgery
Brief Title: The Role Of Noninvasive 320-Row Multidetector Computer Tomography
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 08-0033-BE
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease
Keywords: CAD; CTCA; multidetector computer tomography (MDCT)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Computer tomography coronary angiogram (CTCA) has emerged as a noninvasive alternative to assessing coronary artery luminal disease. Although the use of noninvasive CTCA for the detection of coronary artery disease is on the rise, the current technology of the 64-row multidetector computer tomography (MDCT) is subjected to multiple patient artifacts that can affect image quality.To eliminate these patient related artifacts a more advanced 320-row MDCT was recently developed. The investigators therefore propose that the newly developed 320-MDCT can provide an accurate noninvasive assessment of the severity of coronary artery luminal stenosis as an alternative to an invasive coronary angiogram.

DETAILED DESCRIPTION:
This pilot study consisting of a prospective non-randomized observational trial where a team of surgeon, anesthesiologist, and evaluator are blinded to CTCA results. We hypothesize that the preoperative use of noninvasive computer tomography, with the 320-row MDCT, to visualize the degree of coronary artery stenosis can lead to improved clinical prediction of perioperative cardiac complications.

The 320-row MDCT is based on the 64-row technology with the significant addition of a larger detector capable of scanning the heart within 1 sec or a cardiac cycle, thereby, eliminating patient-related artifacts and may produce higher image quality.13, 14 The scanning time of 5 seconds with the 320-row MDCT is significantly reduced compared to 8-10 seconds for the 64-row MDCT

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years and older
* Able to understand and willing to sign the Informed Consent Form
* Undergoing vascular surgery or intermediate risk surgery (these include intraperitoneal, intrathoracic, carotid endarterectomy , head and neck, orthopedics or prostate) AND
* One or more of the following clinical predictors according to the Revised Cardiac Risk Index:

  1. history of ischemic heart disease (CABG, MI, Stent, positive stress test, Q-waves on ECG)
  2. Diabetes (requiring insulin)
  3. history of congestive heart failure (NYHA I- II)
  4. history of cerebrovascular disease, any of :

     1. history of carotid stenosis
     2. history of ischemic cerebrovascular disease (stroke or TIA)
  5. Aortic or peripheral vascular disease OR
  6. Risk of CAD with 3 or more of the following

     1. Age ≥ 70 years
     2. Hypertension (medicated)
     3. Cholesterol (medicated)
     4. Diabetes (medicated-oral hypoglycemic)
     5. Family history of coronary artery disease

        -

        Exclusion Criteria:
        1. Lack of consent for participation
        2. Pregnancy
        3. History of an allergic response to iodinated contrast medium
        4. History of an allergic response, or other contraindication to beta blockers
        5. eGFR < 45 mL/min
        6. Hemodynamically unstable/compromised
        7. Urgent surgery
        8. Atrial fibrillation > 80 bpm
        9. Uncontrolled tachyarrhythmia
        10. Atrioventricular block (second and third degree)
        11. Moderate to severe aortic stenosis
        12. Not able to hold breath for 5 - 10 seconds
        13. History of multiple myeloma or organ transplant
        14. Severe pulmonary disease including COPD, PAH, asthma
        15. Congestive heart failure presented as NYHA functional class III - IV
        16. Severe anemia
        17. Increased intracranial pressure
        18. Closed angle glaucoma
        19. Absolute contraindication to Nitroglycerin
        20. Presence of medical condition or history that investigator feels would be problematic
        21. Acute myocardial infarction (within 4-6 weeks) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - stable patients undergoing intermediate or high risk elective non-cardiac surgical procedure according to the American Heart Association/American College of Cardiology (AHA/ACC) Guideline for Perioperative Cardiovascular Evaluation for Non-Cardiac Surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-09; Primary Completion 2014-06 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To assess the coronary luminal stenosis for location, number of vessels involved and severity of luminal stenosis using noninvasive CTCA. | CTCA 1-2 hours
  CTCA will be read by a cardiac radiologist blinded to the patients' medical/cardiac history and the results of the stress test. The cardiac radiologist will classify the severity of coronary artery disease according to number of vessels, location and degree of luminal steno-occlusive disease.

SECONDARY OUTCOMES:
Perioperative cardiac complications | In hospital day 0-3, 30 days post surgery and one year
  Non-fatal and fatal cardiac complications will be reviewed day 0- 3 and day 30 post-surgery and one year. Patients who are discharged home will be contacted by telephone by a research assistant for post-operative follow-up. Non-fatal cardiac complications include myocardial infarction, arrythmias, electrocardiogram ischemic changes, cardiac enzymes elevation, symptoms of congestive heart failure and/or angina

CONTACTS AND LOCATIONS:
Overall Officials: Eric You Ten Kong, MD PhD FRCPC, Principal Investigator — Mount Sinai Hospital, University Health Network
Locations (1):
- University Heatlh Network, Mount Sinai, Toronto General Hopsital sites, Toronto, Ontario, Canada